CLINICAL TRIAL: NCT01090557
Title: A Prospective, Pilot Study Measuring Exhaled Nitric Oxide Levels in Infants and Young Children Admitted to the Hospital for Respiratory Syncytial Virus (RSV) or Other Viral Lower Respiratory Tract Infections
Brief Title: Exhaled Nitric Oxide in Respiratory Syncytial Virus (RSV) Bronchiolitis: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Maria Lyn Quintos-Alagheband, MD, Division of Pediatric Critical Care,Winthrop University Hospital
Other Study IDs: 07029
Record Dates: First submitted 2009-10-06; First posted 2010-03-22 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2010-03

CONDITIONS: RSV Infection; Bronchiolitis
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- RSV positive subjects: Subjects admitted to the hospital with Lower respiratory tract Viral infection symptoms from which nasopharyngeal mucous samples are positive for RSV by Direct Fluorescent Antibody technique and/or viral culture
  Interventions: Other: Collection of exhaled breath
- RSV negative subjects: Subjects admitted to the hospital with Lower respiratory tract Viral infection symptoms from which nasopharyngeal mucous samples are negative for RSV by Direct Fluorescent Antibody technique and/or viral culture (usually positive for influenza A & B, parainfluenza, human metapneumovirus or adenovirus)
  Interventions: Other: Collection of exhaled breath
- Control group: Children with same age range, ethnic background, and gender distribution as the study group coming for evaluation in the outpatient setting without evidence of viral infection
  Interventions: Other: Collection of exhaled breath

INTERVENTIONS:
Other: Collection of exhaled breath — balloon collection, via the tidal breathing techniques with uncontrolled flow rate for offline feNO measurement

SUMMARY:
The fraction of exhaled nitric oxide (feNO) in expired air is a reliable measure of airway inflammation. Some research experiments have demonstrated stimulation of nitric oxide production in respiratory epithelial cells infected with RSV.

The principal aims are to determine if the fraction of exhaled nitric oxide (feNO) is elevated in hospitalized pediatric patients with viral lower respiratory illness and to determine if there is a difference in feNO level between RSV and non-RSV infection.

NO may play a role in the association between RSV, airway reactivity, and airway inflammation.

This is a prospective, pilot study that will noninvasively measure feNO in children 0-4 years of age admitted to Winthrop University Hospital, as well as controls (children in the same age range without respiratory conditions and who are well enough to perform the test). Hospitalized children will be tested for RSV (enzyme immunoassay (EIA) & DFA) and via direct fluorescent antigen technique (DFA) for influenza A & B, parainfluenza, human metapneumovirus and adenovirus.

Method of feNO measurement will utilize the offline options for preschool children & infants appropriate for age as described in the 2005 Joint Statement of the American Thoracic Society & the European Respiratory Society when discussing tidal breathing techniques with uncontrolled flow rate Offline exhaled air can be collected via a mouthpiece or a face mask connected to a non-re-breathing valve that allows inspiration of NO-free air from an NO-inert reservoir to avoid contamination by ambient NO. Exhaled breath samples are collected into an NO-inert bag fitted with the expiratory port once a stable breathing pattern is present.

The results of all 3 groups will be compared: control, RSV positive and RSV negative samples.

ELIGIBILITY:
Inclusion Criteria:

* Admitted subjects with diagnosis of bronchiolitis, viral pneumonia or other significant respiratory viral infection

Exclusion Criteria:

* asthma/RAD
* recurrent wheezing
* "recurrent bronchiolitis"
* allergic rhinitis
* atopy
* chronic lung disease
* hypertension
* heart failure
* pulmonary hypertension
* primary ciliary dyskinesia
* bronchiectasis
* alveolitis
* lung transplant rejection
* pulmonary sarcoidosis
* chronic cough (i.e. greater four weeks)
* systemic sclerosis
* hypersensitivity
* cystic fibrosis
* HIV
* sickle cell anemia
* cardiac pulmonary bypass
* liver cirrhosis
* alpha-1 anti-trypsin disease
* interstitial lung

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The parents of children admitted to WUH with a diagnosis of lower respiratory tract viral illness (LRTVI) will be offered the opportunity to participate
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Difference in feNO level between RSV and non-RSV infection in hospitalized pediatric patients with viral lower respiratory illness as well as with control subjects | 2 years

SECONDARY OUTCOMES:
FeNO levels correlate with the severity of respiratory symptoms in children with acute viral respiratory illness | 2 years
FeNO levels in viral respiratory illness will vary with steroid use | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Quintos-Alagheband, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS recommendations for standardized procedures for the online and offline measurement of exhaled lower respiratory nitric oxide and nasal nitric oxide, 2005. Am J Respir Crit Care Med. 2005 Apr 15;171(8):912-30. doi: 10.1164/rccm.200406-710ST. No abstract available. PMID 15817806
- [Background] Baraldi E, de Jongste JC; European Respiratory Society/American Thoracic Society (ERS/ATS) Task Force. Measurement of exhaled nitric oxide in children, 2001. Eur Respir J. 2002 Jul;20(1):223-37. doi: 10.1183/09031936.02.00293102. PMID 12166573
- [Background] Gentile DA, Doyle WJ, Belenky S, Ranck H, Angelini B, Skoner DP. Nasal and oral nitric oxide levels during experimental respiratory syncytial virus infection of adults. Acta Otolaryngol. 2002 Jan;122(1):61-6. doi: 10.1080/00016480252775751. PMID 11876601
- [Background] Ricciardolo FL, Sterk PJ, Gaston B, Folkerts G. Nitric oxide in health and disease of the respiratory system. Physiol Rev. 2004 Jul;84(3):731-65. doi: 10.1152/physrev.00034.2003. PMID 15269335
- [Background] Kao YJ, Piedra PA, Larsen GL, Colasurdo GN. Induction and regulation of nitric oxide synthase in airway epithelial cells by respiratory syncytial virus. Am J Respir Crit Care Med. 2001 Feb;163(2):532-9. doi: 10.1164/ajrccm.163.2.9912068. PMID 11179135
- [Background] Baraldi E, Dario C, Ongaro R, Scollo M, Azzolin NM, Panza N, Paganini N, Zacchello F. Exhaled nitric oxide concentrations during treatment of wheezing exacerbation in infants and young children. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 1):1284-8. doi: 10.1164/ajrccm.159.4.9807084. PMID 10194178